CLINICAL TRIAL: NCT06220851
Title: Correlation Between Handgrip Strength and Air Trapping in Patients with Stable Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Associate Professor, Thammasat University
Other Study IDs: MTU-EC-IM-0-209/65
Record Dates: First submitted 2024-01-12; First posted 2024-01-24 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; handgrip strength; air trapping; lung volume; correlation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COPD: COPD patients aged 40 years or older with a postbronchodilator ratio of forced expiratory volume at one second (FEV1) to forced vital capacity (FVC) <0.7.
  Interventions: Diagnostic Test: Handgrip strength

INTERVENTIONS:
Diagnostic Test: Handgrip strength — Handgrip strength will be measured by 3 efforts.

SUMMARY:
The goal of this observational study is to investigate the relationship between handgrip strength and air trapping in patients with chronic obstructive pulmonary disease (COPD). The main question it aims to answer is:

• Is handgrip strength correlated with air trapping in COPD patients? Participants will perform handgrip strength test and lung volume measurement.

DETAILED DESCRIPTION:
This is a cross-sectional study in COPD patients. COPD patients aged 40 years or older were included. Handgrip strength test and lung volume measurement will be tested in each patient. Handgrip strength will be measured using a hand dynamometer. Lung volume will be assessed using a body plethysmograph.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Postbronchodilator FEV1/FVC <0.7
* >10 pack-year smoking history

Exclusion Criteria:

* COPD exacerbation within 3 months
* Inability to perform handgrip strength test or lung volume measurement

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients aged 40 years or older who are confirmed diagnosis by spirometry (postbronchodilator FEV1/FVC <0.7) and smoking history 10 pack-years or more.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Correlation between handgrip strength and air trapping in COPD patients | At day 1 of the study
  This correlation will be reported as correlation coefficient (R).

SECONDARY OUTCOMES:
The best cutoff value of handgrip strength for predicting air trapping in COPD patients | At day 1 of the study
  The best cutoff value will be determined by the area under the Receiver Operator Characteristic curve (ROC).

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University Faculty of Medicine, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) and documents will be available for sharing immediately after publication for a period of 2 years.
Supporting Information: Study Protocol, SAP